CLINICAL TRIAL: NCT03207347
Title: A Phase II Trial of the PARP Inhibitor, Niraparib, in BAP1 and Other DNA Damage Response (DDR) Pathway Deficient Neoplasms (UF-STO-ETI-001)
Brief Title: A Trial of Niraparib in BAP1 and Other DNA Damage Response (DDR) Deficient Neoplasms (UF-STO-ETI-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-STO-ETI-001; IRB201701827 -A (Other: University of Florida); OCR15732 (Other: Universiy of Florida)
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Mesothelioma; Uveal Melanoma; Renal Cell Carcinoma; Cholangiocarcinoma
Keywords: BAP1; niraparib; DNA repair; PARP inhibitor; homologous repair deficiency; renal cell carcinoma; cholangiocarcinoma; mesothelioma; uveal melanoma
MeSH Terms: conditions — Mesothelioma; Uveal Melanoma; Carcinoma, Renal Cell; Cholangiocarcinoma | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: Patients in both cohorts will receive niraparib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): This cohort will enroll patients with mesothelioma, uveal melanoma, renal cell carcinoma (clear cell type), and cholangiocarcinoma.
  Interventions: Drug: Niraparib
- Cohort B (Experimental): This cohort will enroll patients whose tumors have a known DNA damage response mutation in any of the following genes: ARID1A, ATM, ATR, BACH1 (BRIP1), BAP1, BARD1, BLM, CHEK1, CHEK2, CDK2, CDK4, ERCC, FAM175A, FEN1, IDH1, IDH2, MRE11A, NBN (NBS1), PALB2, POLD1, PRKDC (DNA-PK) PTEN, RAD50, RAD51, RAD52, RAD54, RPA1, SLX4, WRN, or XRCC. This cohort is open to patients with any type of malignancy (except prostate).
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Patients will take 300 mg of niraparib orally once daily each day of a 28 day cycle.
  Other Names: Zejula

SUMMARY:
This open-label, non-randomized study will investigate the use of niraparib in patients with tumors known to have mutations in BAP1 and other select DNA damage response pathway genes.

DETAILED DESCRIPTION:
BAP1 is an ubiquitin ligase that is critical in helping to regulate the cell cycle, cellular differentiation, and cell death. This protein is also intimately involved with DNA double-strand break repair. Germline mutations in the BAP1 gene are associated with a hereditary cancer syndrome that increases the risk of uveal melanoma, mesothelioma and renal cell carcinoma. PARP is another protein that is crucial in DNA repair and enables continued cell replication and survival. It is hypothesized that PARP inhibition with niraparib will result in significant cytoreduction in patient tumors with mutations in BAP1 and other components of the DNA damage response pathway through synthetic lethality. Synthetic lethality is the inhibition of a gene that a cell relies on to compensate for the loss of another gene, resulting in the cell's demise.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed clinical diagnosis of incurable cancer
* Confirmed diagnosis of uveal melanoma, mesothelioma, renal cell carcinoma (clear cell subtype), or cholangiocarcinoma (Cohort A only)
* Known DNA damage repair mutation including any one of the following: ARID1A, ATM, ATR, BACH1 (BRIP1), BAP1, BARD1, BLM, CHEK1, CHEK2, CDK2, CDK4, ERCC, FAM175A, FEN1, IDH1, IDH2, MRE11A, NBN (NBS1), PALB2, POLD1, PRKDC (DNA-PK) PTEN, RAD50, RAD51, RAD52, RAD54, RPA1, SLX4, WRN, or XRCC. Only CLIA certified next generation sequencing (NGS) assays are acceptable. Variants of unknown significance (VUS) will be allowed to enroll on study. (Cohort B only)
* Prior treatment with standard systemic therapy (must have exhausted or declined all known and currently approved effective life prolonging therapies)
* Must have formalin-fixed paraffin embedded (FFPE) tissue available for research purposes. Tissue must have been obtained within the last 3 years from a core or excisional biopsy.
* Measurable disease by RECIST (v 1.1) criteria
* Adequate organ function
* ECOG Performance Status of 0-1
* Life expectancy ≥ 12 weeks
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to the first dose AND be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 180 days after the last dose of study drug to minimize the risk of pregnancy.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 180 days following the last dose of study drug. In addition, men must not donate sperm during niraparib therapy and for 180 days after receiving the last dose of niraparib.
* Subjects must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Subjects receiving oral corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
* If a new biopsy is needed for diagnostic reasons, the biopsy must be performed from a tumor site that is not the only site of measurable disease.

Exclusion Criteria:

* Prior exposure to PARP inhibitors
* Subject has received or is planning to receive live vaccines within 30 days prior to the first dose of oral treatment and while participating in the trial
* Known BRCA1 or BRCA2 mutation
* Pathologic diagnosis of prostate cancer as the cancer to be treated in cohort B
* Simultaneous enrollment in any other interventional clinical trial
* Major surgery ≤ 3 weeks of study enrollment (Subject must have recovered from any effects of any major sugery.)
* Investigational therapy ≤ 4 weeks of first day of dosing of study drug
* Radiotherapy to > 20% of the bone marrow within 4 weeks of the first dose of study drug
* Known hypersensitivity to the components of niraparib or the excipients
* Platelet or red blood cell transfusion ≤ 4 weeks of first dose of study drug
* Colony-stimulating factors within 4 weeks prior to starting protocol therapy
* More than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treatment physician and approved by the PI] may be included).
* Known, active symptomatic brain or leptomeningeal metastases
* Subject has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Known history of myelodysplastic syndrome or acute myeloid leukemia
* Females or males of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for at least 180 days after the last dose of study drug.
* Females who are pregnant or breastfeeding
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician or study PI.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas George, MD, FACP, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] George TJ, Lee JH, DeRemer DL, Hosein PJ, Staal S, Markham MJ, Jones D, Daily KC, Chatzkel JA, Ramnaraign BH, Close JL, Ezenwajiaku N, Murphy MC, Allegra CJ, Rogers S, Zhang Z, Li D, Srinivasan G, Shaheen M, Hromas R. Phase II Trial of the PARP Inhibitor, Niraparib, in BAP1 and Other DNA Damage Response Pathway-Deficient Neoplasms. JCO Precis Oncol. 2024 Dec;8:e2400406. doi: 10.1200/PO-24-00406. Epub 2024 Dec 3. PMID 39626160

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort B (Closed to Enrollment): This cohort will enroll patients whose tumors have a known DNA damage response mutation in any of the following genes: ARID1A, ATM, ATR, BACH1 (BRIP1), BAP1, BARD1, BLM, CHEK1, CHEK2, CDK2, CDK4, ERCC, FAM175A, FEN1, IDH1, IDH2, MRE11A, NBN (NBS1), PALB2, POLD1, PRKDC (DNA-PK) PTEN, RAD50, RAD51, RAD52, RAD54, RPA1, SLX4, WRN, or XRCC. This cohort is open to patients with any type of malignancy (except prostate).
  Niraparib: Patients will take 300 mg of niraparib orally once daily each day of a 28 day cycle.
Period: Overall Study
Arm/Group | Cohort A | Cohort B (Closed to Enrollment)
Started | 23 | 14
Completed | 23 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B (Closed to Enrollment) | Total
Number analyzed (Participants) | 23 | 14 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 16 | 6 | 22
Age, Continuous [Mean (Full Range); unit: years] | 65.57 [39 to 86] | 61.43 [33 to 73] | 64.00 [33 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 13 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 14 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 21 | 13 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 14 | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Determine the objective response rate (ORR), which is defined as the percentage of subjects achieving a best overall response of partial or complete response (according to RECIST v1.1 criteria) from the start of the treatment until disease progression/recurrence or 30 days after the end of treatment, whichever occurs first. Per RECIST v1.1 criteria, a partial response is defined as a 30% or more decrease in the sum of the largest diameters of the target lesions. Per RECIST v1.1 criteria, a complete response is defined as the disappearance of target lesions (lymph nodes identified as lesions must have reduction in short axis to <10 mm).
Time Frame: 1 year
Population: The analysis population for both cohorts only includes those subjects with at least one RECIST response assessment at the end of treatment. 6 subjects (5 subjects in Cohort A and 1 subject in Cohort B) did not have at lease one RECIST response assessment at the end of treatment and are not included in the analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 18 | 13
percentage of subjects | 5.6 [0.1 to 27.3] | 0 [0 to 0]

2. Secondary Outcome: Progression-Free Survival
Description: Determine the median progression-free survival. Progression-free survival is defined as the duration of time from study entry to time of progression or death or the date of last contact, whichever occurs first. Progression is defined by RECIST v1.1 criteria and is defined as an increase of at least 20% in the sum of the largest diameters of target lesions and/or the appearance of new lesions.
Time Frame: 8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 23 | 14
months | 2.1 [1.8 to 9.1] | 7.2 [1.8 to 12.5]

3. Secondary Outcome: Progression-Free Survival Rate at 3 Months
Description: Determine the progression-free survival rate at 3 months after study entry in each cohort. This is the percentage of subjects that both have not had disease progression and are alive 3 months after study entry. Disease progression is defined by RECIST v1.1 criteria and is defined as an increase of at least 20% in the sum of the largest diameters of target lesions and/or the appearance of new lesions.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 23 | 14
percentage of subjects | 43 [23 to 62] | 64 [34 to 83]

4. Secondary Outcome: Progression-Free Survival Rate at 6 Months
Description: Determine the progression-free survival rate at 6 months after study entry in each cohort. This is the percentage of subjects that both have not had disease progression and are alive 6 months after study entry. Progression is defined by RECIST v1.1 criteria and is defined as an increase of at least 20% in the sum of the largest diameters of target lesions and/or the appearance of new lesions.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 23 | 14
percentage of subjects | 39 [20 to 58] | 57 [28 to 78]

5. Secondary Outcome: Overall Survival
Description: Estimate the median overall survival. Overall survival is defined as the duration of time from date of study entry until date of death or date of last contact.
Time Frame: 10 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 23 | 14
months | 9.1 [2.0 to 13.0] | 7.2 [2.9 to 15.5]

ADVERSE EVENTS:
Time Frame: Serious adverse events and adverse events of special interest were collected, at a minimum, from the time of informed consent until 90 days after the last dose of niraparib. All other adverse events were collected, at a minimum, from the time of informed consent until 30 days after the last dose of niraparib. Adverse events were collected for a maximum of 911 days.
Description: All adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator. Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 23/23 | 14/14
Serious Adverse Events (participants affected / at risk) | 8/23 | 7/14
Other Adverse Events (participants affected / at risk) | 23/23 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=23) | Cohort B (N=14)
Lung infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Unknown infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=23) | Cohort B (N=14)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Alanine aminotransferase increased (Investigations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 7 | 0
Anemia (Blood and lymphatic system disorders) | 7 | 2
Anorexia (Metabolism and nutrition disorders) | 9 | 7
Anxiety (Psychiatric disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Enlarged groin lymph nodes (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Creatinine increased (Investigations) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dizziness (Nervous system disorders) | 5 | 1
Dry eye (Eye disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Edema limbs (General disorders) | 1 | 2
Esophageal ulcer (Gastrointestinal disorders) | 1 | 0
Itchy eyes (Eye disorders) | 1 | 0
Fatigue (General disorders) | 17 | 8
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Fever (General disorders) | 0 | 4
Flu like symptoms (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Oral petechia (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Transaminitis (Hepatobiliary disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Stomach virus (Infections and infestations) | 0 | 1
Inflammation and yellow discharge around insertion site nephrostomy (Infections and infestations) | 0 | 1
Cold (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 12 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Platelet count decreased (Investigations) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Right ureteral stenosis (Renal and urinary disorders) | 0 | 1
Sinus pain (Nervous system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin tear (Skin and subcutaneous tissue disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Weight loss (Investigations) | 6 | 4
White blood cell decreased (Investigations) | 1 | 1
Diabetes type 2 (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03207347/Prot_SAP_000.pdf